CLINICAL TRIAL: NCT04516421
Title: Protein Supplementation Intervention for Improving Muscle Mass and Physical Performance in Older People With Sarcopenia: A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Protein Supplementation Intervention for Improving Muscle Mass and Physical Performance in Older People With Sarcopenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Asia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: JWang20-CF01
Record Dates: First submitted 2020-08-10; First posted 2020-08-18 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Sarcopenia
Keywords: older people; sarcopenia; handgrip strength; muscle mass
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: Then eligible participants is invited to attend this randomized, double-blind, placebo-controlled,2-parallel-group trial, and concealed allocation and intention-to-treat (ITT) analysis were applied, and randomly assigned to the experimental and control group in the ratio of 1:1 for the 12-week trial. and intervention.
Who Masked: Participant, Care Provider
Masking Description: After random assignment, the external researcher newly assigned a subject ID to each participant. All other study personnel and participants remained blinded to the identity codes throughout the course of the study. When participants withdrew from or completed the study, researchers were provided with the participants' identities, and the participants were told what supplement they had received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will receive a 12-weeks intervention, with each day a pack of supplementation containing 14g protein, 0.6g fat, 7g carbohydrate, 4.4 g BCAA , 2.4g glutamate, 0.5g arginine and 0.4g taurine with 90 kcal/pack (Affix Health, Taiwan Branch).
  Interventions: Dietary Supplement: Protein supplementation
- Control (Placebo) group (Placebo Comparator): The control (placebo) group will receive a 12-week oat drink, with each day a pack of oat tea containing 1.5g protein, 0.5g fat, 0.1g carbohydrate with 8.3kcal/pack (Zhan Xuan, Co. Ltd., Taiwan).
  Interventions: Dietary Supplement: Placebo oat drink

INTERVENTIONS:
Dietary Supplement: Protein supplementation — The experimental group contained 14g protein, 0.6g fat, 7g carbohydrate, 4.4 g BCAA , 2.4g glutamate, 0.5g arginine and 0.4g taurine with 90 kcal/pack (Affix Health, Taiwan Branch).
  Arms: Experimental group
Dietary Supplement: Placebo oat drink — placebo oat drink contained 1.5g protein, 0.5g fat, 0.1g carbohydrate with 8.3kcal/pack (Zhan Xuan, Co. Ltd., Taiwan).
  Arms: Control (Placebo) group

SUMMARY:
Background: Declines in muscle mass and strength are expected with aging, but physical inactivity and low protein intake have been suggested as risk factors of sarcopenia. So far, lifestyle interventions, especially exercise and nutritional supplementation, prevail as mainstays of treatment for sarcopenia.

Objective: To explore the effect and benefits of protein supplementation on the improvement of muscle mass and physical performance in older people with sarcopenia.

Design: A randomized, double-blind, placebo-controlled clinical trial. Methods: Participants aged 65-95y who meet the following criteria will be invited: (1) muscle mass: bioimpedance, <7.0 kg/m² (male) and <5.7 kg/m² (female), (2) handgrip strength: <28 kg (male) and <18 kg (female), and (3) low physical performance: 6-m gait Speed <1.0 m/s. Study participants will be randomly assigned to two groups. The experimental group will receive a 12-week intervention with【protein (14g)+ BCAA(4.4g)】 drink per day, while the parallel control group will receive a placebo oat drink per day.

Participants in the control group will be asked to maintain participants' usual diet and physical activity. There are 3 time-points to measure outcomes and observe other required information, at week 0(baseline), 6 and 12.

DETAILED DESCRIPTION:
Background: Sarcopenia is defined as an abnormal loss of muscle mass and strength. Declines in muscle mass and strength are expected with aging, but physical inactivity and low protein intake have been suggested as risk factors of sarcopenia. Recently, Taiwan is known as the fastest-aging nation in the world, and the prevalence of sarcopenia has been reported as 3.9-7.3%; even more 9-64% in Dr. Chen's study. So far, lifestyle interventions, especially exercise and nutritional supplementation, prevail as mainstays of treatment for sarcopenia.

Objective: To explore the effect and benefits of protein supplementation on the improvement of muscle mass and physical performance in older people with sarcopenia.

Study design: A randomized, double-blind, placebo-controlled clinical trial which will be conducted between September and November, 2020.

Participants: The study will be conducted in Keelung, Taiwan. A total of 9 day-care centers, including 180 over 65 years of residents, will be invited to participate the study via telephone calls.

Eligible participants will be invited to attend this randomized, double-blind, placebo-controlled, 2-parallel-groups trial, and will be randomly assigned to the experimental and control groups with 1:1 ratio.

Intervention: The intervention period will be 12 weeks. The control group will receive 150c.c placebo oat drink (1.5g protein, 0.5g fat, 0.1g carbohydrate each pack, Zhan Xuan Co. Ltd., Taiwan) per day, five days per week, while the experimental group will receive 150c.c protein supplementation drink (14g protein, 0.6g fat, 7g carbohydrate, 4.4 g BCAA , 2.4g glutamate, 0.5g arginine and 0.4g taurine each pack, Affix Health, Taiwan Branch) per day, five days per week.

Supplementation in the experimental group contains 90 kcal/d and the placebo oat drink contains 8.3kcal/d. Participants in the control group will be asked to maintain participants' usual diet and physical activity. There are 3 time-points to measure outcomes and observe other required information, at week 0(baseline), 6 and 12.

Sample size calculation: Referring to the setting in a published paper that gave a sample size of 30 participants/group, a sample size of 40 participants in each group is considered in the study, by considering potential dropouts.

Random assignment and blinding: An independent external researcher prepared a computer generated cluster random sampling. After random assignment, the external researcher newly assigned a subject ID to each participant. All other study personnel and participants remained blinded to the identity codes throughout the course of the study. When participants withdrew from or completed the study, researchers were provided with the participants' identities, and the participants were told what supplement participants had received.

Ethical approval: The study was approved by Taipei Hospital Human Trial Committee of the Ministry of Health and Welfare. All participants were assured that data collected from participants would be strictly conﬁdential, and the physical condition and safety were given priority. Investigators conducted intervention only after obtaining participants ethical approval (registration number: TH-IRB-00190046). Anyone who feel uncomfortable during the study will be allowed to quit immediately with no any restriction.

Study measurement: Kihon Checklist, MNA, GDS-SF, SPPB, IADL, MMSE, handgrip, 6m gait speed, (SMI), SF-12 questionnaire and Tw-FROP-Com.

Statistical methods: Statistical analysis was conducted using the IBM SPSS software (version 22, IBM Corporation, New York, NY). An intention-to-treat analysis was performed. (1) Descriptive statistics: describe the distribution of category variables by number and percentage, and the mean and standard deviations describe the distribution of continuous variables. (2) Inference statistics: chi-square: to verify whether the pre-measured category variants between the experimental group and the control group are homogeneous. ANOVA: Check whether the continuous variables measured between the experimental group and the control group are homogeneous. Generalized estimating equations (GEE) with interactions of time and group in the models will be conducted to evaluate the intervention effect. A two-sided p-value < 0.05 is considered statistically signiﬁcant.

ELIGIBILITY:
Inclusion Criteria:

* 65-95 years old
* can communicate in Mandarin or Taiwanese language
* sacorpenia (basing on criteria of Asian Working Group for Sarcopenia )

Exclusion Criteria:

* with liver or kidney disease
* stent in body.

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-08-24 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Skeletal muscle mass index ("change" is being assessed) | The change is assessed from week 0 (baseline) to week 12
  Bioimpedance is adopted to assess sarcopenia. Therefore, Skeletal muscle mass index is measured by bioimpedance( using the In body instrument Model 230) and means ASM/H²((sum of lean muscle mass in upper and lower limb divided by square of body height). Skeletal muscle mass index is used with a cut-off value of 7 kg/m² in men, and 5.4 kg/m² in women according to the AWGS 2020.

SECONDARY OUTCOMES:
Hand-grip strength ("change" is being assessed) | The change is assessed from week 0 (baseline) to week 12
  The maximal hand grip strength is measured using a Camry (Model:EH101) hand dynamometer. The investigator will demonstrate how to use the dynamometer, then participants will be asked to press for 3 to 5 seconds on the grip using the greatest possible force. The measurement is repeated after a 30-second rest. Both hands will be measured separately and the highest score is registered. The cut-off value of hand-grip is <28 kg for men and <18 kg for women according to the AWGS 2019..
Gait speed ("change" is being assessed) | The change is assessed from week 0 (baseline) to week 12
  Gait speed means measurement of 6 meters walking speed. The cut-off value of gait speed is <1.0 m/s according to the AWGS 2019.

OTHER OUTCOMES:
Short Physical Performance Battery ("change" is being assessed) | The change is assessed from week 0 (baseline) to week 12
  The SPPB includes usual walking speed 4 m, five chair-stands test, and balance test. A score (scale: 0-4) is assigned to performance on time to rise five times from a seated position, standing balance, and 4-m walking velocity. participants receive a score of 0 for unable to complete each task. Summing the three individual categorical scores, a summary performance score is created for each participant (range: 0-12), with higher scores indicating better body function. In the walking test, the participants could use a cane, a walker, or other walking aid but the aid of another person. The cut-off value is ≦9 according to the AWGS 2019.
Instrumental Activities of Daily Living ("change" is being assessed) | The change is assessed from week 0 (baseline) to week 12
  There are eight domains of function measured with the Lawton IADL scale. Women are scored on all 8 areas of function; historically, for men, the areas of food preparation, housekeeping, laundering are excluded. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women, and 0 through 5 for men. There are 3 of 5 ( Shopping,Mode of Transportation, Food Preparation,Laundry and Housekeeping) in need of assistance is mild inability.
Mini-Mental State Examination ("change" is being assessed) | The change is assessed from week 0 (baseline) to week 12
  The MMSE scores may be used to classify the severity of cognitive impairment or to document serial change in dementia participants. A full score of 30 indicates that the higher score means better cognitive function. The following four cut-off levels should be employed to classify the severity of cognitive impairment: no cognitive impairment 24-30; mild cognitive impairment 19-23; moderate cognitive impairment 10-18; and severe cognitive impairment ≤9.
Falls Risk for Older People Community setting-Taiwan Version ("change" is being assessed) | The change is assessed from week 0 (baseline) to week 12
  The tool consists of 13 factors being rated, most on a graded 0-3 scale, and thus ranges from 0 to 60. A higher score indicates a higher risk. The fall risk score can be divided into 3 levels: high(19- 60), medium(12- 18) and light( 0 - 11).
Medical Outcome Study Short Form-12 ("change" is being assessed) | The change is assessed from week 0 (baseline) to week 12
  The SF-12 which provides information on mental and physical health status is a shortened version of the SF-36. The SF-12 uses the same eight domains as the SF-36. The total score is from 0 to 8. The higher the score, the better quality of life.
Geriatric depression scale-short form ("change" is being assessed) | The change is assessed from week 0 (baseline) to week 12
  GDS-SF is a measure designed to explore depression associated with the elderly. There are a total of 15 self-made scales of questions, each of which respondents only have to answer yes or no.The total score is 15 , the cutoff values is 5, more than 5 means depression symptoms, the higher score , the higher degree of depression.
Kihon Checklist-Chinese ("change" is being assessed) | The change is assessed from week 0 (baseline) to week 12
  A tool for measuring the degree of frailty of the elderly, There were 25 test assessments in the scale, and if there were more than five, the weaker the participantes were.
Taiwan-Mini Nutritional Assessment ("change" is being assessed) | The change is assessed from week 0 (baseline) to week 12
  It is a nutritional assessment scale suitable for Taiwan's elderly over 65years old with severe malnutrition. The total score is 14. The higher score means more better. The score of 12-14 means normality, 8-11 means malnutrition-risk, and less and equal 7 means malnutrition.

CONTACTS AND LOCATIONS:
Overall Officials: Chang, Principal Investigator — Ching Kuo Institute of Management and Health, Keelung, Taiwan
Locations (3):
- Taiwan (3):
  - Keelung Hospital Daycare Center, Ministry of Health and Welfare, Keelung
  - Keelung First Daycare Center, Keelung
  - Keelung Second Daycare Center, Keelung

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen LK, Woo J, Assantachai P, Auyeung TW, Chou MY, Iijima K, Jang HC, Kang L, Kim M, Kim S, Kojima T, Kuzuya M, Lee JSW, Lee SY, Lee WJ, Lee Y, Liang CK, Lim JY, Lim WS, Peng LN, Sugimoto K, Tanaka T, Won CW, Yamada M, Zhang T, Akishita M, Arai H. Asian Working Group for Sarcopenia: 2019 Consensus Update on Sarcopenia Diagnosis and Treatment. J Am Med Dir Assoc. 2020 Mar;21(3):300-307.e2. doi: 10.1016/j.jamda.2019.12.012. Epub 2020 Feb 4. PMID 32033882